CLINICAL TRIAL: NCT02824380
Title: Pharmacokinetics/ Pharmacodynamics and Safety of DA-4001 in Healthy Male Subjects With Androgenic Alopecia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA4001_AGAP_I
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

ARMS (2):
- Sequence A (Experimental): Period 1: DA-4001 H(High dose) Period 2: DA-4001 L(Low dose)
  Interventions: Drug: DA-4001 H; Drug: DA-4001 L
- Sequence B (Experimental): Period 1: DA-4001 L(Low dose) Period 2: DA-4001 H(High dose)
  Interventions: Drug: DA-4001 H; Drug: DA-4001 L

INTERVENTIONS:
Drug: DA-4001 H — 5% minoxidil / high dose of finasteride
Drug: DA-4001 L — 5% minoxidil / low dose of finasteride

SUMMARY:
An Open-label, Randomized, Multiple-dose, Crossover Study to Evaluate the Pharmacokinetics/ Pharmacodynamics and Safety of DA-4001 in Healthy Male Subjects with Androgenic Alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged between 19 and 65 years, clinically healthy
* BMI between 18.5kg/m2 and 27kg/m2
* Clinical history of Androgenic Alopecia

Exclusion Criteria:

* Subject has any dermatological disorders of the scalp
* Subject has a history of hair transplants, hair weaves
* Subject has hypersensitivity to previously prescribed minoxidil or finasteride
* Subject who is considered inappropriate to participate in the study due to any conditions including screening results at the investigator's discretion

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Css,max(Maximum steady state concentration) of Finasteride(ng/mL) | day1, 6: before administration, day7: before administration and 0.5, 1, 2, 3, 4, 6, 8, 12, 24h after administration
AUCtau(Area under the plasma concentration versus time curve) of Finasteride (ng·hr/mL) | day1, 6: before administration, day7: before administration and 0.5, 1, 2, 3, 4, 6, 8, 12, 24h after administration
Change from baseline of testosterone and DHT(ng/mL) | day1: before administration, day7: before administration and 6, 12, 24h after administration

SECONDARY OUTCOMES:
Tss,max(Time to reach maximal serum concentrations at steady state)of Finasteride(hr) | day1, 6: before administration, day7: before administration and 0.5, 1, 2, 3, 4, 6, 8, 12, 24h after administration
Css,min(Minimum steady state concentration)of Finasteride(ng/mL) | day1, 6: before administration, day7: before administration and 0.5, 1, 2, 3, 4, 6, 8, 12, 24h after administration
t1/2β(Elimination Half-life) of Finasteride(hr) | day1, 6: before administration, day7: before administration and 0.5, 1, 2, 3, 4, 6, 8, 12, 24h after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea